CLINICAL TRIAL: NCT07016568
Title: Temporary Aortic Occlusion With the Abdominal Tourniquet for Refractory Postpartum Haemorrhage: A Proof-of-Concept Study in a War-Affected Region
Acronym: TAOAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LLC UkrMedGroup (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024/EC/128094
Record Dates: First submitted 2025-06-04; First posted 2025-06-11 (Actual); Results first posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Postpartum Haemorrhage (PPH)
Keywords: uterine atony; postpartum haemorrhage; Emergency Obstetric Care; Aortic Compression
MeSH Terms: conditions — Postpartum Hemorrhage; Uterine Inertia

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-arm, open-label proof-of-concept study. All eligible participants will receive the investigational intervention (AAJT-S device) as an adjunct to standard care for severe postpartum hemorrhage unresponsive to uterotonics and balloon tamponade. No comparator or control group is included. The study is designed to evaluate feasibility, safety, and preliminary clinical outcomes in a conflict-affected, resource-limited setting.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AAJT-S Device Intervention Arm (Experimental): Participants in this arm will receive standard postpartum hemorrhage (PPH) management followed by application of the Abdominal Aortic and Junctional Tourniquet - Stabilized (AAJT-S) device if bleeding remains uncontrolled after uterotonics and uterine balloon tamponade. The device will be applied to the upper abdomen and inflated to 250 mmHg to achieve temporary aortic occlusion for up to 60 minutes. The intervention is intended to temporize bleeding while definitive surgical treatment and blood transfusion are arranged.
  Interventions: Device: Abdominal Aortic and Junctional Tourniquet - Stabilized (AAJT-S)

INTERVENTIONS:
Device: Abdominal Aortic and Junctional Tourniquet - Stabilized (AAJT-S) — The AAJT-S is a non-invasive, externally applied medical device designed to achieve temporary occlusion of the abdominal aorta and inferior vena cava by inflating a pneumatic bladder to 250 mmHg. In this study, the device will be used as a temporizing measure for patients with severe postpartum hemorrhage unresponsive to standard uterotonics and balloon tamponade. The device will be applied horizontally over the upper abdomen and inflated using a built-in pressure gauge. The intended effect is to reduce pelvic blood flow and allow time for mobilization of surgical resources and blood transfusion. Maximum application time will not exceed 60 minutes, in accordance with established safety guidelines.

SUMMARY:
The purpose of this study is to evaluate whether a medical device called the Abdominal Aortic and Junctional Tourniquet - Stabilized (AAJT-S) can safely and effectively temporarily stop severe bleeding after childbirth (known as postpartum hemorrhage) when standard treatments fail. The main question the study aims to answer is: Can the AAJT-S device temporarily control life-threatening postpartum bleeding long enough to allow doctors to prepare for surgery and other definitive treatment?

DETAILED DESCRIPTION:
This prospective, open-label, non-randomized, proof-of-concept study will assess the feasibility, safety, and preliminary clinical effectiveness of the Abdominal Aortic and Junctional Tourniquet - Stabilized (AAJT-S) device as a temporizing measure for severe postpartum hemorrhage (PPH) due to uterine atony that is unresponsive to standard first-line therapies. The study will be conducted in a tertiary referral center in Zaporizhzhia, Ukraine, located in a conflict-affected region with limited access to timely surgical intervention and blood products.

Eligible participants will be adult postpartum patients (≥18 years) who develop primary PPH with blood loss exceeding 1,000 mL and who fail to respond to pharmacologic uterotonics and balloon tamponade. Patients with hemorrhage due to trauma, coagulopathy, or retained placental tissue will be excluded.

Once standard management protocols are exhausted and eligibility is confirmed, the AAJT-S device will be deployed over the upper abdomen and inflated to 250 mmHg to achieve temporary occlusion of the abdominal aorta and inferior vena cava. The device is intended to reduce pelvic blood flow and thereby control hemorrhage during the critical window required to mobilize a surgical team, arrange blood transfusion, and secure anesthesia.

The device will remain in place for a maximum of 60 minutes, consistent with published safety guidelines. Clinical endpoints will include time to bleeding control, hemodynamic stabilization, need for additional surgical intervention, and total blood loss. Safety endpoints will include thrombotic events, ischemic injury, infections, and any other adverse events related to device use.

Data will be collected prospectively, including demographic characteristics, obstetric history, timing and duration of interventions, and perioperative outcomes. Descriptive statistics will be used to summarize findings, with no formal hypothesis testing due to the pilot nature of the study.

All participants will receive routine inpatient follow-up, and longer-term outcomes will be assessed via scheduled in-person visits and structured telephone interviews at 6 and 12 months postpartum to evaluate for delayed complications and maternal recovery. The study is designed to generate preliminary data for further exploration of the AAJT-S device as a potential emergency tool for PPH management in resource-limited and crisis settings.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Clinical diagnosis of postpartum hemorrhage (PPH) refractory to uterotonics and intrauterine balloon tamponade
* Estimated blood loss greater than 1,000 mL
* Oral informed consent provided prior to device application

Exclusion Criteria:

* Patients with postpartum bleeding as a result of trauma, retained placenta or coagulopathy were excluded

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Self-identified females who are biologically capable of pregnancy and childbirth are eligible to participate. The study includes individuals assigned female at birth with a functioning uterus who have delivered vaginally and experienced postpartum hemorrhage. Participation is limited to those with physiologic ability to undergo the obstetric processes being studied.
Enrollment: 4 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Viktor Oshovskyy, DMSc, PhD, MD, Principal Investigator — pirhospr@gmail.com
Locations (1):
- Olexandrivska Hospital, Zaporizhzhia, Ukraine

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the small sample size and the sensitive nature of the clinical context, including emergency obstetric care in a war-affected setting. Additional ethical and regulatory considerations related to patient privacy and consent limit the possibility of external data sharing.

REFERENCES:
- [Background] Soltan MH, Sadek RR. Experience managing postpartum hemorrhage at Minia University Maternity Hospital, Egypt: no mortality using external aortic compression. J Obstet Gynaecol Res. 2011 Nov;37(11):1557-63. doi: 10.1111/j.1447-0756.2011.01574.x. Epub 2011 Jun 16. PMID 21676082
- [Background] Soltan MH, Faragallah MF, Mosabah MH, Al-Adawy AR. External aortic compression device: the first aid for postpartum hemorrhage control. J Obstet Gynaecol Res. 2009 Jun;35(3):453-8. doi: 10.1111/j.1447-0756.2008.00975.x. PMID 19527382
- [Background] Kheirabadi BS, Dubick MA. Safe duration of Abdominal Aortic and Junctional Tourniquet application. J Trauma Acute Care Surg. 2019 Sep;87(3):740-741. doi: 10.1097/TA.0000000000002231. No abstract available. PMID 30768561
- [Background] Nieto-Calvache AJ, Palacios-Jaraquemada JM, Aryananda RA, Basanta N, Cininta N, Rivera-Torres LF, Bautista E, Hussein AM. External aortic compression: buying time to save lives in obstetric hemorrhage. Am J Obstet Gynecol. 2025 Feb;232(2):239-241. doi: 10.1016/j.ajog.2024.09.017. Epub 2024 Sep 18. No abstract available. PMID 39304012
- [Background] Riley DP, Burgess RW. External abdominal aortic compression: a study of a resuscitation manoeuvre for postpartum haemorrhage. Anaesth Intensive Care. 1994 Oct;22(5):571-5. doi: 10.1177/0310057X9402200512. PMID 7818062
- [Background] Nieto-Calvache AJ, Palacios Jaraquemada JM, Basanta N, Aryananda RA, Sinisterra-Diaz SE, Rodriguez F, Hidalgo Cardona A, Messa Bryon A. Internal manual compression of the aorta-an effective way to temporarily control pelvic bleeding in obstetrical hemorrhage. Am J Obstet Gynecol. 2022 Jul;227(1):96-97. doi: 10.1016/j.ajog.2022.02.040. Epub 2022 Mar 4. PMID 35248574
- [Background] Khan M, Jeyanathan J, Smith JE. Novel use for the abdominal tourniquet in the management of postpartum haemorrhage. J R Army Med Corps. 2018 Nov;164(6):463. doi: 10.1136/jramc-2018-000953. Epub 2018 Apr 6. No abstract available. PMID 29626141
- See also: Information about The Abdominal Aortic and Junctional Tourniquet - Stabilized (AAJT-S) — https://www.narescue.com/abdominal-aortic-and-junctional-tourniquet-stablized-aajt-s.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at Olexandrivska Hospital (Zaporizhzhia, Ukraine) between December 2024 and April 2025. Recruitment was based on clinical diagnosis of refractory postpartum hemorrhage due to uterine atony, and all participants provided oral informed consent.
Pre-assignment Details: All enrolled participants (N=4) met the eligibility criteria and were assigned to the intervention arm. No screening failures, exclusions, or withdrawals occurred prior to device application.
Groups:
- Experimental: AAJT-S Device Intervention Arm: Participants in this arm received standard postpartum hemorrhage (PPH) management followed by application of the Abdominal Aortic and Junctional Tourniquet - Stabilized (AAJT-S) device if bleeding remains uncontrolled after uterotonics and uterine balloon tamponade. The device was applied to the upper abdomen and inflated to 250 mmHg to achieve temporary aortic occlusion for up to 60 minutes. The intervention was intended to temporize bleeding while definitive surgical treatment and blood transfusion are arranged.
Period: Overall Study
Arm/Group | Experimental: AAJT-S Device Intervention Arm
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental: AAJT-S Device Intervention Arm
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Region of Enrollment [Number; unit: Participants]
  Ukraine | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Parity [Mean (Standard Deviation); unit: Births] — Number of previous deliveries (including both vaginal and cesarean births) prior to the index pregnancy.
  Births | 2.5 (1.7)
Estimated Blood Loss Prior to AAJT-S Application [Mean (Full Range); unit: ml] — Volume of blood loss assessed by gravimetric methods before placement of the AAJT-S device.
  ml | 1125 [1030 to 1200]

OUTCOME MEASURES:

1. Primary Outcome: Time to Bleeding Control After AAJT-S Device Application
Description: Defined as the time (in minutes) from inflation of the AAJT-S device to visible cessation of external vaginal bleeding in patients with severe postpartum hemorrhage due to uterine atony. Bleeding control will be determined by visual clinical assessment by the attending provider. This measure evaluates the immediate effectiveness of the intervention in stopping hemorrhage and buying time for definitive surgical management or transfusion.
Time Frame: Within 10 minutes of AAJT-S device application
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | AAJT-S Device Intervention Arm
Number analyzed (Participants) | 4
Minutes | 2 (0.01)

2. Primary Outcome: Total Measured Blood Loss (Pre- and Post-intervention)
Description: Sum of blood loss (in mL), measured by pad/towel weights after AAJT-S use until definitive hemostasis.
Time Frame: From onset of PPH until bleeding is definitively controlled (typically within 1-6 hours)
Measure: Mean (Full Range); unit: ml
Arm/Group | AAJT-S Device Intervention Arm
Number analyzed (Participants) | 4
ml | 1425 [1150 to 1800]

3. Primary Outcome: Incidence of Device-related Complications
Description: Includes thrombotic events, ischemic injury, skin necrosis, or technical malfunction during/after AAJT-S use.
Time Frame: From device application through hospital discharge (up to 7 days)
Measure: Count of Participants; unit: Participants
Arm/Group | AAJT-S Device Intervention Arm
Number analyzed (Participants) | 4
Participants | 0

4. Secondary Outcome: Hemodynamic Stabilization Time
Description: Time from device inflation to achievement of target blood pressure (SBP ≥90 mmHg) and pulse <110 bpm.
Time Frame: First 60 minutes after AAJT-S application
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | AAJT-S Device Intervention Arm
Number analyzed (Participants) | 4
Minutes | 31.25 (6.29)

5. Secondary Outcome: Long-term Maternal Recovery Status
Description: Assessed via follow-up calls and scheduled ultrasound visits at 6 weeks postpartum, including return to normal activity, presence of chronic pain, or menstrual abnormalities.
Time Frame: At 6 weeks postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | AAJT-S Device Intervention Arm
Number analyzed (Participants) | 4
Participants | 4

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, up to 12 weeks
Arm/Group | AAJT-S Device Intervention Arm
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
* Small sample size prevents generalizability.
* No control group.
* Estimates of blood loss may be subject to observer bias.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-11-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT07016568/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT07016568/SAP_001.pdf